CLINICAL TRIAL: NCT03016130
Title: A Phase III, Randomized, Clinical Trial Comparing Two Diets in Patients Undergoing Hematopoietic Stem Cell Transplant (HSCT) or Remission Induction Chemotherapy for Acute Leukemia and Myelodysplastic Syndrome (UF-BMT-LDND-101)
Brief Title: Comparing Two Diets in Patients Undergoing HSCT or Remission Induction Chemo for Acute Leukemia and MDS (UF-BMT-LDND-101)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis determined that study reached a safety stopping rule
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201700581; UF-BMT-LDND-101 (Other: University of Florida); OCR15632 (Other: UF OnCore); UF-HEM-007 (Other: University of Florida)
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: leukemia; myelodysplastic; myeloid; lymphoblastic; diet; infection; hematopoietic; stem cell; transplant
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Infections | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberalized Hospital Diet (Diet A) (Active Comparator): Diet A would include fresh fruits and/or fresh vegetables in a liberalized hospital diet, and subjects will be encouraged to eat at least one daily serving of fresh fruits and/or vegetables.
  Interventions: Other: Diet
- Neutropenic Diet (Diet B) (Active Comparator): Diet B is the hospital neutropenic diet.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Diet Intervention: Subjects will undergo stratified randomization to account for the heterogeneous population, to receive one of the two diets: liberalized hospital diet (Diet A) or a neutropenic diet (Diet B).

SUMMARY:
This is an open-label, two-arm, phase III non-inferiority trial to evaluate the safety of a liberalized hospital diet inclusive of fresh fruits and vegetables to a neutropenic diet in patients with prolonged neutropenia. Both cohorts and diets will adhere to the hygiene and common sense advice listed in the FDA-endorsed food safety guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing treatment for hematologic malignancies or HSCT as outlined below:
* Underlying diagnosis for non-HSCT patients:
* Acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) receiving induction or reinduction chemotherapy; OR
* Acute lymphoblastic leukemia (ALL) receiving an intensive induction chemotherapy (e.g., HyperCVAD±R, CALGB9251, Larsons protocol) with an expected duration of neutropenia of ≥7 days; OR
* Allogeneic or autologous HSCT for any indication. For patients undergoing reduced intensity conditioning, only those regimens in which the expected neutropenia is ≥ 7 days are permitted and the patient must reside in the hospital
* Expected duration of neutropenia of ≥ 7 days

Exclusion Criteria:

* Use of anti infectives for treatment of active systemic infections within 7 days prior to initiation of study diet
* Untreated major infection at presentation
* Patients with uncontrolled invasive fungal infection (defined as those who have not completed at least 6 weeks of treatment; or who are symptomatic with two CT scans, at least 1 week apart showing uncontrolled disease at the time of initiation of study diet)
* Uncontrolled HIV, Hepatitis B and C infection
* Receipt of nutrition via enteral tube or total parenteral nutrition at the time of enrollment
* Patients unwilling to eat fresh fruit and/or vegetables
* Planned management of neutropenia in the outpatient setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Incidence of major infections | 1 year
  The primary objective of the trial is to compare the incidence of major infections in subjects undergoing HSCT or receiving induction chemotherapy for acute leukemia with prolonged neutropenia (less than or equal to 7 days) who are receiving either Diet A or Diet B.

SECONDARY OUTCOMES:
Incidence of infections in each diet group | 1 year
  This secondary objective of the trial is to compare the impact of diet on severe infections including: septic shock, bloodstream infection, invasive fungal infection, upper respiratory infection, infectious & non-infectious pneumonia, C. difficile infection, Vancomycin-resistant & -sensitive enterococcal colonization, Vancomycin-resistant & -sensitive enterococcal infections, febrile neutropenia, typhlitis, lower tract respiratory viral infections, infection-related mortality, and admission to the ICU.
Admission frequency | 1 year
  This secondary objective of the trial will examine the admission frequency to the intensive care unit (ICU).
Compliance | 1 year
  This secondary objective of the trial will evaluate the degree of compliance to each diet from the time of initiation of the diet intervention until either the Absolute Neutrophil Count (ANC) is equal to or less than 500/mm3, the subject is discharged from the hospital, the subject is transferred from the unit, or after 30 days of ANC less than 500/mm3.
Patient-Generated Subjective Global Assessment (PG-SGA) | 1 year
  This secondary objective of the trial will evaluate the impact of each diet on nutritional status as assessed by PG-SGA.
Incidence of mucositis | 1 year
  This secondary objective of the trial will evaluate the impact of mucositis on dietary intake.
Symptom incidence | 1 year
  This secondary objective of the trial is to compare symptoms between diets using the MDASI tool.
Quality of life (QoL) | 1 year
  This secondary objective of the trial is to compare the QoL between diets as assessed by FACT-G.
Overall survival (OS) | 1 year
  This secondary objective of the trial is to evaluate OS from 1 year following randomization
Progression free survival (PFS) | 1 year
  This secondary objective of the trial is to evaluate PFS from 1 year following randomization
Incidence of graft vs.host disease (GVHD) | 1 year
  This secondary objective of the trial is to evaluate the incidence of GVHD in allogeneic HSCT subjects only.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crispen, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Wingard JR, Lee JH, Li D, Al-Mansour Z, Farhadfar N, Hsu J, Hiemenz J, Dean EA, Brown R, Trikha G, Schulz JN, Cline CL, Leather H, Sugrue MW, Dahl WJ, McGee KH, Leggett A, Kelly DL. Randomized Noninferiority Trial of a Liberalized Diet Versus the Neutropenic Diet in Hematopoietic Stem-Cell Transplant Patients and Patients With Acute Leukemia. J Clin Oncol. 2026 Feb;44(4):300-310. doi: 10.1200/JCO-25-00889. Epub 2025 Dec 17. PMID 41406403